CLINICAL TRIAL: NCT00007969
Title: A Phase 1/2 Uncontrolled, Open Label Study Of Photodynamic Vaccination In Patients With Stage III/IV Malignant Melanoma
Brief Title: Photodynamic Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: QLT Inc. (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068358; QLT-VFI-PDV-01; QLT-PHO-VFI-PDV-01
Record Dates: First submitted 2001-01-06; First posted 2004-03-11 (Estimated); Last update posted 2013-11-06 (Estimated); Status verified 2008-08

CONDITIONS: Melanoma (Skin)
Keywords: stage III melanoma; stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — detox adjuvant; Verteporfin

INTERVENTIONS:
Biological: Detox-B adjuvant
Drug: verteporfin

SUMMARY:
RATIONALE: Photodynamic therapy uses light and drugs that make cancer cells more sensitive to light to kill tumor cells. Photodynamic therapy may be effective in treating melanoma.

PURPOSE: Phase I/II trial to study the effectiveness of photodynamic therapy in treating patients who have stage III or stage IV melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of photodynamic therapy with verteporfin and Detox-B adjuvant in patients with stage III or IV melanoma. II. Determine the clinical response in patients treated with this regimen. III. Determine whether this regimen induces systemic cellular and humoral immune responses to melanoma antigens in these patients. IV. Determine the ablation of cutaneous tumors in patients treated with this regimen.

OUTLINE: This is a multicenter study. Patients undergo photodynamic therapy with verteporfin and Detox-B adjuvant. Treatment repeats every 2 weeks for a total of 3 courses, each to a different melanoma lesion. Both non-treated and treated tumors are measured prior to study and at months 2, 4, and 6. Immune profile is also assessed prior to study and at months 2, 4, and 6.

PROJECTED ACCRUAL: A total of 30 patients will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Diagnosis of stage III or IV melanoma At least 3 cutaneous tumors for treatment (treatment tumors) AND 1-7 additional cutaneous, visceral, or lymph node tumors for response assessment (marker tumors) Treatment tumors must be on trunk, arms, or legs AND be 1.0-3.6 cm in longest dimension Measurable disease by calipers or CT scan No CNS metastases by CT scan

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: ECOG 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 2,500/mm3 Neutrophil count at least 1,000/mm3 Platelet count at least 50,000/mm3 Hemoglobin at least 9 g/dL Hematocrit at least 27% Hepatic: Bilirubin no greater than 2 times upper limit of normal (ULN) AST/ALT no greater than 2 times ULN Alkaline phosphatase no greater than 2.5 times ULN Renal: Creatinine no greater than 2 times ULN

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy or immunotherapy No concurrent biologic therapy Chemotherapy: At least 4 weeks since prior chemotherapy No concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy No concurrent radiotherapy Surgery: No concurrent surgical removal of melanoma lesions designated for treatment or response assessment Other: No other concurrent therapy for melanoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-10

CONTACTS AND LOCATIONS:
Overall Officials: Graeme R. Boniface, PhD, Study Chair — QLT Inc.
Locations (6):
- United States (6):
  - University of Colorado Cancer Center, Denver, Colorado
  - Mount Sinai Comprehensive Cancer Center at Aventura, Aventura, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Missouri Baptist Cancer Center, St Louis, Missouri
  - University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania